CLINICAL TRIAL: NCT02424669
Title: Neuroinflammation in Amyotrophic Lateral Sclerosis - Mechanisms and Therapeutic Perspectives: a Translational Pilot Study Among ALS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2014-19; RCAPHM15_0132 (Registry Identifier: Assistance Publique Hôpitaux Marseille)
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Blood Specimen Collection

ARMS (3):
- recently diagnosed ALS patients (Experimental)
  Interventions: Other: ALS Functional rating Scale-revised (ALS FRS-R); Other: slow vital capacity; Other: Blood sample; Other: Cerebrospinal Fluid (CSF) sample
- not recently diagnosed ALS patients (Experimental)
  Interventions: Other: ALS Functional rating Scale-revised (ALS FRS-R); Other: slow vital capacity; Other: Blood sample; Other: Cerebrospinal Fluid (CSF) sample
- patients with peripheral neuropathy, recently diagnosed (Active Comparator)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: ALS Functional rating Scale-revised (ALS FRS-R)
  Arms: not recently diagnosed ALS patients; recently diagnosed ALS patients
Other: slow vital capacity
  Arms: not recently diagnosed ALS patients; recently diagnosed ALS patients
Other: Blood sample
Other: Cerebrospinal Fluid (CSF) sample
  Arms: not recently diagnosed ALS patients; recently diagnosed ALS patients

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is the most common motor neuron diseases. It is considered as a rare disease with a prevalence of about 8 per 100,000 persons. Initiating in mid-life by progressive paralysis, it evolves rapidly into a generalized muscle wasting that leads irrevocably to death within 2 or 5 years of clinical onset.

Since there is no cure for ALS, the management of the disease is supportive and palliative. Riluzole is the only drug that has been shown to extend survival by about three months. The identification of biomarkers sensitive to the progression of the disease might enhance the diagnostic and provide new drug targets.

Dysfunction of the immune system is a pathological hallmark of ALS. Increased levels of interferon gamma (IFNgamma) were found in the serum and cerebrospinal fluid (CSF) of ALS patients. However, the cell origin as well as the pathogenic influence of this peripheral source of IFNg is unknown. Thus, IFNgamma might have a role in the pathogenic process of ALS and might be a potential biomarker of the disease.

ELIGIBILITY:
Inclusion Criteria:

Group 1 and Group 2:

* with sporadic ALS (without family history), recently diagnosed (onset of first symptoms < 24 months) group 1, not recently diagnosed (onset of first symptoms > 24 months) group 2
* Who meet the laboratory-supported probable, probable or definite form of ALS according to the El Escorial criteria
* Suffering from the spinal form of ALS

Group 3:

- with an inflammatory peripheral neuropathy, or a non inflammatory peripheral neuropathy, recently diagnosed

Exclusion Criteria:

* Familial form of ALS
* Bulbar form and respiratory onset form of ALS
* Subjects with a clinically significant history of unstable or severe cardiac, oncologic, hepatic or renal disease, or other medically significant illness.
* Subjects with significant cognitive impairment, clinical dementia, or psychiatric illness.
* Female of childbearing potential (apart of patient using adequate contraceptive measures), pregnant or breast feeding
* Suspected inability to complete the study follow-up (foreign workers, transient visitors, tourists or any others for whom follow-up evaluation is not assured)
* Participation in any other clinical study within 30 days prior to the Screening Visit
* Persons deprived of freedom by judicial or administrative decision, hospitalized without their consent or for other reasons than the research, under legal protection or unable to express their consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
ALS Functional rating Scale-revised (ALS FRS-R) score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France